CLINICAL TRIAL: NCT02564588
Title: A 12-week, Randomized, Double-blind, Parallel-group, Placebo Controlled, Flexibly Dosed, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Dasotraline in Adults With Moderate to Severe Binge Eating Disorder
Brief Title: Dasotraline Binge Eating Disorder Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP360-221
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dasotraline (Experimental): Dasotraline 4, 6, 8 mg
  Interventions: Drug: Dasotraline
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dasotraline — Dasotraline 4, 6, 8mg flexibly dosed once daily
  Arms: Dasotraline
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
Evaluate the efficacy of flexibly-dosed dasotraline compared with placebo in adults with moderate to severe Binge Eating Disorder (BED)

DETAILED DESCRIPTION:
This is a randomized, double blind, parallel group, multicenter, outpatient study evaluating the efficacy and safety of flexibly-dosed dasotraline in adults with BED using dasotraline (4, 6, and 8 mg/day) versus placebo over a 12 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 55 years of age, inclusive, at time of informed consent.
* Subject meets the following DSM 5 criteria for a diagnosis of BED. An episode of binge eating is characterized by both:
* Eating an amount of food larger than what most people would eat, in a discrete period of time (eg, 2 hours)
* Sense of lack of control over eating episode
* Binge-eating episodes are associated with ≥ 3 of the following:
* Eating much more rapidly than normal
* Eating until uncomfortably full
* Eating large amounts when not feeling hungry
* Eating alone because of embarrassment
* Feeling disgusted with oneself, guilty afterward
* Binge-eating episodes are also associated with marked distress regarding the episode and not associated with recurrent use of compensatory behavior (eg, bulimia nervosa).
* Diagnosis is confirmed based on the eating-disorders module of the SCID, clinician review of subject diaries, and the EDE Q.
* Subject has a BED diagnosis including at least 2 binge eating days a week for at least 6 months prior to screening.
* Subject's BED is of at least moderate severity.
* Subject has a negative breath alcohol test and a negative urine drug screen (UDS) for any illicit drug.
* Female subject must have a negative serum pregnancy test at screening; females who are post-menopausal (defined as at least 12 months of spontaneous amenorrhea) and those who have undergone hysterectomy or bilateral oophorectomy will be exempted from the pregnancy test.
* Female subject of childbearing potential and male subject with female partner of childbearing potential must agree to use an effective and medically acceptable form of birth control throughout the study period. Note: Continued use of an effective and medically acceptable form of birth control is recommended for 30 days after study completion.
* Subject must be able to comply with study drug administration and adhere to protocol requirements.

Subject can read well enough to understand the informed consent form and other subject materials.

Exclusion Criteria:

* Subject has body weight index (BMI) of 18 kg/m2or less or greater than 45 kg/m2.
* Subject has a lifetime history or current symptoms of bulimia nervosa or anorexia nervosa.
* Subject has started psychotherapy (eg, supportive psychotherapy, cognitive behavior therapy, interpersonal therapy) within 3 months prior to screening. Note: Subjects receiving stable ongoing psychotherapy for longer than 3 months are permitted to enroll.
* Subject is participating in a formal weight loss program (eg, Weight Watchers®) within 3 months prior to screening.
* Subject has used a psychostimulant or mood stabilizer within the 3 months prior to screening.
* Subject has used any medications for the treatment of binge eating, other eating disorders, obesity, or weight gain or any other medication that could result in weight gain or weight loss including over-the-counter and herbal products within the 3 months prior to screening.
* Subject has a lifetime history of psychotic disorder, bipolar disorder, hypomania, dementia, or ADHD as defined by the DSM 5 criteria.
* Subject has a history of moderate to severe depression based on investigator's judgment within the 6 months prior to screening or is currently taking or has taken any medication for depression during the 3 months prior to screening.
* Subject has a history of substance use disorder including alcohol use disorder (excluding nicotine and caffeine) within the 12 months prior to screening, as defined by the DSM 5 criteria.
* Subject has MADRS score ≥ 18 at screening and Baseline visit.
* Subject is considered a suicide risk or has any previous history of suicide attempt.
* Subject answers "yes" to "suicidal ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C SSRS assessment at screening (in the past month). Subjects who answer "yes" to this question must be referred to the Investigator for follow up evaluation.
* Subject has type I diabetes mellitus or insulin-dependent diabetes mellitus.
* Subject with type II diabetes mellitus has hemoglobin A1c ≥ 6.5% at screening, or has initiated treatment with or changed the dose of a glucose-lowering agent within 3 months prior to screening.
* Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, documented heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems.
* Subject has initiated treatment with or changed the dose of a lipid-lowering medication within the 3 months prior to screening.
* Subject has a history of moderate or severe hypertension that in the investigator's opinion has not been medically stable or has required a change in dosage and/or medication during the 3 months prior to screening.
* Subject has a history of epilepsy, seizures (except childhood febrile seizures), unexplained syncope or other unexplained blackouts (except single incident), or head trauma with loss of consciousness lasting more than 5 minutes, or a history of clinically significant repeated head-traumas without loss of consciousness.
* Subject is female and pregnant or nursing.
* Subject has had bariatric surgery, lap bands, duodenal stents, or other procedures for weight loss.
* Subject has a history of positive test for Hepatitis B surface antigen or Hepatitis C antibody with liver function test results at screening above the upper limit of normal (ULN) for the reference laboratory.
* Subject without a history of positive test for Hepatitis B surface antigen or Hepatitis C antibody has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value ≥ 2 times the ULN at screening.
* Subject has a blood urea nitrogen (BUN) value ≥ 1.5 times the ULN for the reference range, fasting blood glucose ≥ 126 mg/dL (7.0 mmol/L), or hemoglobin A1c ≥ 6.5% at screening.
* Subject is known to have tested positive for human immunodeficiency virus (HIV).
* Subject has a clinically significant abnormality on screening evaluation including physical examination, vital signs, ECG, or laboratory tests that the investigator considers to be inappropriate to allow participation in the study.
* The subject's screening ECG shows a corrected QT interval using Fridericia's formula (QTcF) of ≥ 450 msec for male subjects or ≥ 470 msec for female subjects. Eligibility will be based on the core laboratory ECG interpretation report.
* Subject has any life-time history of abuse or diversion of stimulants.
* Subject has a history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the study drug formulation.
* Subject has enrolled in any Phase 2 or 3 trial of psychostimulants including lisdexamfetamine dimesylate (Vyvanse®) for binge-eating disorder.
* Subject is currently participating or has participated in any clinical trial within the last 90 days or has participated in more than 2 clinical trials within the past year. This includes studies using marketed compounds or devices.
* Subject has previously been enrolled in a clinical trial of dasotraline (SEP 225289).
* Subject is an investigational site staff member or the relative of an investigational site staff member.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 319 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of binge days (defined as days during which at least 1 binge episode occurs) per week to Week 12 | 12 Weeks

SECONDARY OUTCOMES:
Change from baseline in number of binge episodes per week to Weeks 1, 2, 3, 4, 6, 8, 10, and 12 | 12 Weeks
Percent of subjects with a 4-week cessation from binge eating (defined as a 100% reduction for at least 28 consecutive days in the number of binge eating episodes prior to the EOT visit) | 4 weeks
Change from baseline in Clinical Global Impression-Severity (CGI S) score at Weeks 2, 4, 6, 8, 10, and 12 | 12 Weeks
Change from baseline in Eating Disorder Examination Questionnaire Brief Version (EDE Q7) global score and 3 subscale scores (dietary restraint, shape/weight overvaluation, and body dissatisfaction) at Weeks 4, 8, and 12 | 12 Weeks
Change from baseline in Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (Y BOCS BE) total score and subscale scores (obsessions and compulsions) at Weeks 2, 4, 6, 8, 10, and 12 | 12 Weeks
Change from baseline in Sheehan disability Scale (SDS) total score and subscale scores (school/work disability, social life disability, and family life disability at Week 12 | 12 Weeks
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total score at Week 12 | 12 Weeks
Change from baseline in Hamilton Anxiety Rating Scale (HAM A) score at Week 12 | 12 Weeks
Change from baseline in Medical Outcomes Study 12 Item Short Form (SF 12) two component scores (physical component, mental health component) at Week 12 | 12 Weeks
Proportion of binge-eating responders who have ≥ 75% reduction in the number of binge eating episodes from Baseline at Week 12 | 12 weeks
Proportion of binge-eating responders who have ≥ 50% reduction in the number of binge eating episodes from Baseline at Week 12 | 12 Weeks
The incidence of overall AEs, serious AEs (SAEs), and AEs (or SAEs) leading to discontinuations | 12 Weeks
Clinical laboratory evaluations (serum chemistry, hematology, and urinalysis) | 12 Weeks
Clinical evaluations (vital signs, orthostatic effects, and 12 lead ECGs) | 12 Weeks
Frequency and severity of suicidal ideation and suicidal behavior as assessed by the Columbia-suicide severity rating scale (C SSRS) | 12 Weeks
Change and percent change from baseline in body weight at Weeks 1, 2, 3, 4, 6, 8, 10, and 12 | 12 Weeks
Change and percent change from baseline in BMI at Weeks 1, 2, 3, 4, 6, 8, 10, and 12 | 12 Weeks
Change from baseline in a fasting lipid panel (triglycerides, total cholesterol, high-density lipoprotein [HDL] cholesterol, and low-density lipoprotein [LDL] cholesterol) at Weeks 6 and 12 | 12 Weeks
Change from baseline in hemoglobin A1c level at Weeks 6 and 12 | 12 Weeks
Change from baseline in fasting glucose level at Weeks 6 and 12 | 12 Weeks
Change in the symptoms of withdrawal from Week 12/end of treatment (EOT) as measured by: - CSSA scores at Weeks 13, 14, and 15 - DESS scores at Weeks 13, 14, and 15 - HAM A scores at Weeks 13, 14, and 15 - MADRS scores at Weeks 13, 14, and 15. | 3 Weeks
  The change in symptoms of withdrawal is a time frame of 3 weeks after treatment ends (weeks 13, 14, 15)

CONTACTS AND LOCATIONS:
Overall Officials: Dasotraline Medical Director, MD, Study Director — Sunovioin
Locations (43):
- United States (43):
  - Southern California Research, Beverly Hills, California
  - Southwestern Research, Inc., Beverly Hills, California
  - Pharmacology Research Institute, Encino, California
  - Collaborative NeuroScience Network Inc., Garden Grove, California
  - Pharmacology Research Institute, Newport Beach, California
  - PCSD- Feighner Research, San Diego, California
  - Research Across America, Santa Ana, California
  - Lytle and Weiss, PLLC, Denver, Colorado
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Institute of Advanced Medical Research, Alpharetta, Georgia
  - Neurotrials Research, INC., Atlanta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Goldpoint Clinical Research, Inc., Indianapolis, Indiana
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - McLean Hospital, Belmont, Massachusetts
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Princeton Medical Institute, LCC, Princeton, New Jersey
  - Bioscience Research, LLC, Mount Kisco, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Radiant Research, Inc., Akron, Ohio
  - Patient Priority Clinical Sites, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Lindner Center Of Hope, Mason, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Oregon Center for Clinical Investigatons, INC., Portland, Oregon
  - Oregon Center for Clinical Investigatons, INC., Salem, Oregon
  - Lehigh Center For Clinical Research, Allentown, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Furturesearch Trials of Dallas, Dallas, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Psychiatric Medical Associates, Plano, Texas
  - Radiant Research, Inc., Murray, Utah
  - Advanced Research Institute, Ogden, Utah
  - Neuropsychiatric Associates, Woodstock, Vermont
  - NeuroScience, Inc., Herndon, Virginia
  - Summit Research Network (Seattle) LLC, Seattle, Washington

REFERENCES:
- [Derived] McElroy SL, Hudson JI, Grilo CM, Guerdjikova AI, Deng L, Koblan KS, Goldman R, Navia B, Hopkins S, Loebel A. Efficacy and Safety of Dasotraline in Adults With Binge-Eating Disorder: A Randomized, Placebo-Controlled, Flexible-Dose Clinical Trial. J Clin Psychiatry. 2020 Sep 8;81(5):19m13068. doi: 10.4088/JCP.19m13068. PMID 32926604